CLINICAL TRIAL: NCT01062841
Title: Targeted Infection Control Program (TIP) to Reduce Resistant Pathogens and Infections
Brief Title: Targeted Infection Control in Long-term Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Lona Mody, Associate Professor, Internal Medicine, Division of Geriatric and Palliative Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AG032298-01A1
Record Dates: First submitted 2010-02-02; First posted 2010-02-04 (Estimated); Results first posted 2016-09-29 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-08

CONDITIONS: Infection
Keywords: Long-Term Care; Nursing Homes; Infection Control; Multi-drug resistant pathogens; Long-term care residents with in-dwelling devices
MeSH Terms: conditions — Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention: Targeted Infection Control (Active Comparator): Nursing homes allocated to the Intervention Arm will implement a series of new infection control programs.
  Interventions: Behavioral: Targeted Infection Control
- Control (No Intervention): Nursing homes allocated to the control group will continue with their standard infection control procedures. No changes will be made to their practices.

INTERVENTIONS:
Behavioral: Targeted Infection Control — Component 1: Institute enhanced barrier precautions for all NH residents with indwelling devices; active screening for MDROs (monthly) using cultures collected from multiple body sites to identify asymptomatic MDRO carriage in these residents; and dissemination of results to clinical staff and administration.
  Component 2: Structured, active surveillance for infections using standardized definitions in residents with indwelling devices and dissemination of results to clinical staff and administration.
  Component 3: A hand hygiene promotion program. Component 4: A structured educational program pertaining to indwelling device care for healthcare workers.
  Arms: Intervention: Targeted Infection Control

SUMMARY:
This is an interventional study aimed at reducing multi-drug resistance and infections in nursing home (NH) residents. Each year, a staggering 1.5-2.0 million infections occur in NHs. Many of these infections are caused by multiple drug resistant organisms (MDROs) including methicillin-resistant Staphylococcus aureus (MRSA), vancomycin-resistant enterococci (VRE), and multidrug resistant Gram-negative bacilli (R-GNB). Antimicrobial resistance among common bacteria are adversely affecting the clinical course and exponentially increasing healthcare costs. Recognizing a need for action, legislators, policy makers, and consumer groups are advocating for pathogen-based universal preemptive screening for these MDROs, particularly MRSA in hospitals and NHs. However, implementing this sweeping mandate is controversial, costly, reactive, and not based on empirical evidence. It can result in a 10-20-fold increase in the number of NH residents placed in isolation precautions with the potential for reduced attention by healthcare workers, isolation and functional decline. The investigators proposal evaluates a novel focused approach between 'do nothing' and 'search all and destroy' strategies by targeting a subgroup of NH residents with indwelling devices who are at a high risk of acquiring MDROs and infections.

The investigators hypothesize that the investigators targeted infection control program (TIP) will reduce MDRO colonization and infections in NH residents with indwelling devices. This cluster randomized trial will involve 12 NHs; 6 will be randomized to the TIP arm and 6 to the routine care arm. The investigators TIP intervention will include four components.

DETAILED DESCRIPTION:
Component 1: Institute enhanced barrier precautions for all NH residents with indwelling devices; active screening for MDROs (monthly) using cultures collected from multiple body sites to identify asymptomatic MDRO carriage in these residents; and dissemination of results to clinical staff and administration.

Component 2: Structured, active surveillance for infections using standardized definitions in residents with indwelling devices and dissemination of results to clinical staff and administration.

Component 3: A hand hygiene promotion program.

Component 4: A structured educational program pertaining to indwelling device care for healthcare workers.

ELIGIBILITY:
Inclusion Criteria:

* Any short- or long-stay resident with an indwelling urinary catheter or feeding tube for more than 72 hours
* Ability to get informed consent from either the resident or his/her durable power of attorney

Exclusion Criteria:

* Having an indwelling device for less than 72 hours
* Refusal of consent to get surveillance cultures and data collection by the resident or his/her durable power of attorney
* Residents who are receiving end-of-life care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Actual)
Dates: Start 2010-05; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lona Mody, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan and partner nursing homes, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Hutton DW, Krein SL, Saint S, Graves N, Kolli A, Lynem R, Mody L. Economic Evaluation of a Catheter-Associated Urinary Tract Infection Prevention Program in Nursing Homes. J Am Geriatr Soc. 2018 Apr;66(4):742-747. doi: 10.1111/jgs.15316. Epub 2018 Feb 28. PMID 29489017
- [Derived] Cassone M, McNamara SE, Perri MB, Zervos M, Mody L. Impact of Intervention Measures on MRSA Clonal Type and Carriage Site Prevalence. mBio. 2016 Mar 8;7(2):e00218. doi: 10.1128/mBio.00218-16. No abstract available. PMID 26956588
- [Derived] Ismail MD, Luo T, McNamara S, Lansing B, Koo E, Mody L, Foxman B. Long-Term Carriage of Ciprofloxacin-Resistant Escherichia coli Isolates in High-Risk Nursing Home Residents. Infect Control Hosp Epidemiol. 2016 Apr;37(4):440-7. doi: 10.1017/ice.2015.326. Epub 2016 Jan 19. PMID 26782632
- [Derived] Mody L, Krein SL, Saint S, Min LC, Montoya A, Lansing B, McNamara SE, Symons K, Fisch J, Koo E, Rye RA, Galecki A, Kabeto MU, Fitzgerald JT, Olmsted RN, Kauffman CA, Bradley SF. A targeted infection prevention intervention in nursing home residents with indwelling devices: a randomized clinical trial. JAMA Intern Med. 2015 May;175(5):714-23. doi: 10.1001/jamainternmed.2015.132. PMID 25775048

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Residents with an indwelling urinary catheter and/or feeding tube were recruited from 12 nursing homes, May 2010 - April 2013
Groups:
- Intervention: Targeted Infection Control Program: Nursing homes allocated to the Intervention Arm will implement a series of new infection control programs.
  Targeted Infection Control: Component 1: Institute enhanced barrier precautions for all nursing home residents with indwelling devices; active screening for MDRO (multidrug resistant organisms) monthly using cultures collected from multiple body sites to identify asymptomatic MDRO carriage in these residents; and dissemination of results to clinical staff and administration.
  Component 2: Structured, active surveillance for infections using standardized definitions in residents with indwelling devices and dissemination of results to clinical staff and administration.
  Component 3: A hand hygiene promotion program. Component 4: A structured educational program pertaining to indwelling device care for healthcare workers.
- Control: Nursing homes allocated to the control group will continue with their standard infection control procedures. No changes will be made to their practices. Surveillance cultures and data was collected for outcome comparison only.
Period: Overall Study
Arm/Group | Intervention: Targeted Infection Control Program | Control
Started | 203 | 215
Completed | 154 | 162
Not Completed | 49 | 53
Not completed — Indwelling Device Removed | 41 | 48
Not completed — Death | 3 | 5
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Withdrawal by Study | 3 | 0

BASELINE CHARACTERISTICS:
Population: Residents enrolled with >1 follow-up visit
Groups:
- Intervention: Targeted Infection Control Program: Nursing homes allocated to the Intervention Arm will implement a series of new infection control programs.
  Targeted Infection Control: Component 1: Institute enhanced barrier precautions for all nursing home residents with indwelling devices; active screening for MDRO (multidrug resistant organisms) using cultures collected from multiple body sites to identify asymptomatic MDRO carriage in these residents; and dissemination of results to clinical staff and administration.
  Component 2: Structured, active surveillance for infections using standardized definitions in residents with indwelling devices and dissemination of results to clinical staff and administration.
  Component 3: A hand hygiene promotion program. Component 4: A structured educational program pertaining to indwelling device care for healthcare workers.
- Total: Total of all reporting groups
Arm/Group | Intervention: Targeted Infection Control Program | Control | Total
Number analyzed (Participants) | 154 | 162 | 316
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.0 (12.4) | 72.2 (13.5) | 73.1 (12.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 69 | 147
  Male | 76 | 93 | 169
Race/Ethnicity, Customized [Number; unit: participants]
  White Race | 132 | 144 | 276
  Other Race | 22 | 18 | 40
Region of Enrollment [Number; unit: participants]
  United States | 154 | 162 | 316
Charlson's Comorbidity Score [Mean (Standard Deviation); unit: units on a scale] — Charlson's comorbidity score is a weighted index that takes into account the number and seriousness of comorbid disease. It is a classification of comorbid conditions what might alter the risk of mortality in longitudinal studies. 19 conditions are scored with 1, 2, 3, or 6 points. Total Score Range 0 to 37, with increasing scores indicating increasing burden of comorbidity (by increased number of comorbid conditions present, or increased severity of conditions present).
  units on a scale | 2.8 (1.6) | 2.9 (2.1) | 2.9 (1.9)
Physical Self-Maintenance Scale [Mean (Standard Deviation); unit: units on a scale] — Functional disability was assessed using Lawton and Brody's physical self-maintenance scale. Patients are evaluated on their ability to perform six activities of daily living (toileting, feeding, dressing, grooming, bathing, physical ambulation), with 1 = independent, 2 = needs reminders, 3 = needs moderate assistance, 4 = needs extensive assistance, 5 = needs full assistance or resistant to care. The total physical self-maintenance scale ranges from 6 to 30, with increasing scores indicating increasing disability to perform activities of daily living.
  units on a scale | 22.6 (4.1) | 22.1 (4.1) | 22.4 (4.1)
Indwelling Device Use [Number; unit: participants]
  Indwelling Urinary Catheter | 84 | 79 | 163
  Feeding Tube | 46 | 54 | 100
  Both Urinary Catheter and Feeding Tube | 24 | 29 | 53

OUTCOME MEASURES:

1. Primary Outcome: Total Number of MDRO (Multidrug Resistant Organisms) Isolated
Description: Total Number of MDROs isolated across all MDROs and all anatomic sites for all enrolled residents with indwelling devices over the duration of the study period
Time Frame: From enrollment up to 1 year, or until study withdrawal (indwelling device removed, discharged from facility, at resident request, death), or end of study
Population: Residents enrolled with >1 follow-up visit
Measure: Number; unit: Total Number of MDRO isolates
Groups:
- Intervention: Targeted Infection Control Program: Nursing homes allocated to the Intervention Arm will implement a series of new infection control programs.
  Targeted Infection Control: Component 1: Institute enhanced barrier precautions for all NH residents with indwelling devices; active screening for MDROs (monthly) using cultures collected from multiple body sites to identify asymptomatic MDRO carriage in these residents; and dissemination of results to clinical staff and administration.
  Component 2: Structured, active surveillance for infections using standardized definitions in residents with indwelling devices and dissemination of results to clinical staff and administration.
  Component 3: A hand hygiene promotion program. Component 4: A structured educational program pertaining to indwelling device care for healthcare workers.
Arm/Group | Intervention: Targeted Infection Control Program | Control
Number analyzed (Participants) | 154 | 162
Total Number of MDRO isolates | 1299 | 1732
Statistical Analysis 1: Comparison: Intervention: Targeted Infection Control Program vs Control; A mixed-effects multilevel Poisson regression model was used to predict MDRO prevalence density as a function of the intervention (primary outcome), including facility as a random effect and offset by the number of anatomic sites sampled. Because we expected participants colonized at baseline to have a greater likelihood of subsequent colonization, we included participant-level baseline MDRO colonization as a fixed effect; Test type: Superiority or Other; p < 0.05, Regression, Poisson — The model was adjusted for participant-specific covariates (participant-level baseline colonization with the specific MDRO, age, sex, race, and length of stay before enrollment), and NH quality ratings; Rate Ratio = 0.77, 95% CI 2-sided [0.62 to 0.94]

2. Secondary Outcome: Number of First Incident Urinary Catheter-associated Urinary Tract Infections
Time Frame: as for outcome 1
Population: Participants with only a urinary catheter present and >1 follow-up visit
Measure: Number; unit: Number of First CAUTI
Units Other Than Participants: Device-Days
Arm/Group | Intervention: Targeted Infection Control Program | Control
Number analyzed (Participants) | 86 | 80
Number analyzed (Device-Days) | 5982 | 4292
Number of First CAUTI | 31 | 43
Statistical Analysis 1: Comparison: Intervention: Targeted Infection Control Program vs Control; A Cox proportional hazards model using the cluster option with robust standard errors was used to predict time to the first and recurrent infections, adjusting for participant-level and facility-level covariates; Test type: Superiority or Other; p = 0.04, Regression, Cox; Cox Proportional Hazard = 0.54, 95% CI 2-sided [0.30 to 0.97]

3. Primary Outcome: Total Number of MRSA (Methicillin Resistant Staphylococcus Aureus) Isolated
Time Frame: as for outcome 1
Population: Participants with >1 follow-up visit
Measure: Number; unit: Total Number of MRSA isolates
Arm/Group | Intervention: Targeted Infection Control Program | Control
Number analyzed (Participants) | 154 | 162
Total Number of MRSA isolates | 254 | 323
Statistical Analysis 1: Comparison: Intervention: Targeted Infection Control Program vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.05, Regression, Poisson — [p-value comment as in outcome 1, analysis 1]; Rate Ratio = 0.78, 95% CI 2-sided [0.64 to 0.96]

4. Primary Outcome: Total Number of VRE (Vancomycin Resistant Enterococci) Isolated
Time Frame: as for outcome 1
Population: Participants with >1 follow-up visit
Measure: Number; unit: Total Number of VRE isolates
Arm/Group | Intervention: Targeted Infection Control Program | Control
Number analyzed (Participants) | 154 | 162
Total Number of VRE isolates | 122 | 162
Statistical Analysis 1: Comparison: Intervention: Targeted Infection Control Program vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p > 0.05, Regression, Poisson — [p-value comment as in outcome 1, analysis 1]; Rate Ratio = 1.20, 95% CI 2-sided [0.82 to 1.75]

5. Primary Outcome: Total Number of Ceftazidime-resistant GNB (Gram-negative Bacilli) Isolated
Time Frame: as for outcome 1
Population: Participants with >1 follow-up visit
Measure: Number; unit: Total Number of Ceftazidime-RGNB isolate
Arm/Group | Intervention: Targeted Infection Control Program | Control
Number analyzed (Participants) | 154 | 162
Total Number of Ceftazidime-RGNB isolate | 185 | 295
Statistical Analysis 1: Comparison: Intervention: Targeted Infection Control Program vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p > 0.05, Regression, Poisson — [p-value comment as in outcome 1, analysis 1]; Rate Ratio = 0.94, 95% CI 2-sided [0.61 to 1.44]

6. Primary Outcome: Total Number of Ciprofloxacin-resistant GNB (Gram-negative Bacilli) Isolated
Time Frame: as for outcome 1
Population: Participants with >1 follow-up visit
Measure: Number; unit: Total Number of Ciprofloxacin-RGNB
Arm/Group | Intervention: Targeted Infection Control Program | Control
Number analyzed (Participants) | 154 | 162
Total Number of Ciprofloxacin-RGNB | 738 | 952
Statistical Analysis 1: Comparison: Intervention: Targeted Infection Control Program vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.05, Regression, Poisson — [p-value comment as in outcome 1, analysis 1]; Rate Ratio = 0.75, 95% CI 2-sided [0.58 to 0.97]

7. Secondary Outcome: Number of All (First and Recurrent) Incident Urinary Catheter-associated Urinary Tract Infections
Time Frame: as for outcome 1
Population: Participants with only an indwelling urinary catheter present and >1 follow-up visit
Measure: Number; unit: Number of CAUTI
Units Other Than Participants: Device-days
Arm/Group | Intervention: Targeted Infection Control Program | Control
Number analyzed (Participants) | 86 | 80
Number analyzed (Device-days) | 9413 | 8118
Number of CAUTI | 56 | 75

8. Secondary Outcome: Number of Incident Feeding Tube-associated Skin and Soft Tissue Infections
Time Frame: as for outcome 1
Population: Participants with an indwelling feeding tube present (PEG tube), and had >1 follow-up visit
Measure: Number; unit: Numer of feeding-tube SSTIs
Units Other Than Participants: Device-days
Arm/Group | Intervention: Targeted Infection Control Program | Control
Number analyzed (Participants) | 55 | 63
Number analyzed (Device-days) | 5635 | 5062
Numer of feeding-tube SSTIs | 4 | 3
Statistical Analysis 1: Comparison: Intervention: Targeted Infection Control Program vs Control; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.92, Regression, Cox; Cox Proportional Hazard = 1.09, 95% CI 2-sided [0.22 to 5.45]

9. Secondary Outcome: Number of Incident Feeding-tube Associated Pneumonias
Time Frame: as for outcome 1
Population: Participants with indwelling feeding tube present (PEG tube), and had >1 follow-up visit
Measure: Number; unit: Number of feeding-tube associated pneu
Units Other Than Participants: Device-days
Arm/Group | Intervention: Targeted Infection Control Program | Control
Number analyzed (Participants) | 55 | 63
Number analyzed (Device-days) | 5635 | 5062
Number of feeding-tube associated pneu | 10 | 8
Statistical Analysis 1: Comparison: Intervention: Targeted Infection Control Program vs Control; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.34, Regression, Cox; Cox Proportional Hazard = 1.83, 95% CI 2-sided [0.53 to 6.31]

10. Secondary Outcome: Total Number of Residents With New MRSA (Methicillin Resistant Staphylococcus Aureus) Acquisition
Time Frame: as for outcome 1
Population: Participants with >1 follow-up visit, and were at-risk to acquire new MRSA colonization (not colonized at baseline)
Measure: Number; unit: Number of Residents with New MRSA
Units Other Than Participants: Device-days at Risk
Arm/Group | Intervention: Targeted Infection Control Program | Control
Number analyzed (Participants) | 154 | 162
Number analyzed (Device-days at Risk) | 8722 | 7115
Number of Residents with New MRSA | 54 | 56
Statistical Analysis 1: Comparison: Intervention: Targeted Infection Control Program vs Control; A Cox proportional hazards model was used to evaluate the effect of this intervention on an individual's risk of new MDRO acquisition, defined as the number of residents with new acquisitions per 1000 device-days at risk after adjusting for resident-level and facility-level covariates, as well as clustering by facility. Residents colonized with the specific MDRO at baseline were excluded from these analyses; Test type: Superiority or Other; p = 0.01, Regression, Cox; Cox Proportional Hazard = 0.78, 95% CI 2-sided [0.65 to 0.95]

11. Secondary Outcome: Total Number of Residents With New VRE (Vancomycin Resistant Enterococci) Acquisition
Time Frame: as for outcome 1
Population: Participants with > 1 follow-up visit, and who were at-risk to acquire a new VRE colonization (not colonized at baseline)
Measure: Number; unit: Number of Residents with New VRE
Units Other Than Participants: Device-days at Risk
Arm/Group | Intervention: Targeted Infection Control Program | Control
Number analyzed (Participants) | 154 | 162
Number analyzed (Device-days at Risk) | 12756 | 11070
Number of Residents with New VRE | 22 | 26
Statistical Analysis 1: Comparison: Intervention: Targeted Infection Control Program vs Control; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.61, Regression, Cox; Cox Proportional Hazard = 0.85, 95% CI 2-sided [0.45 to 1.60]

12. Secondary Outcome: Total Number of Residents With New Resistant GNB (Ceftazidime or Ciprofloxacin Gram-negative Bacilli) Acquisition
Time Frame: as for outcome 1
Population: Participants with >1 follow-up visit, and who were at-risk to acquire a new R-GNB colonization (not colonized at baseline)
Measure: Number; unit: Number of Residents with New R-GNB
Units Other Than Participants: Device-days at Risk
Arm/Group | Intervention: Targeted Infection Control Program | Control
Number analyzed (Participants) | 154 | 162
Number analyzed (Device-days at Risk) | 7524 | 5685
Number of Residents with New R-GNB | 42 | 35
Statistical Analysis 1: Comparison: Intervention: Targeted Infection Control Program vs Control; Test type: Superiority or Other; p = 0.59, Regression, Cox; Cox Proportional Hazard = 0.90, 95% CI 2-sided [0.60 to 1.33]

ADVERSE EVENTS:
Time Frame: From enrollment up to 1 year, or until study withdrawal (indwelling device removed, discharged from facility, at resident request, death), or end of study
Description: Adverse Events that were Definitely related, Probably related, Possibly related to the study were captured.
  Adverse Events may include: Death, Inpatient hospitalization or prolongation of existing hospitalization, A persistent or significant disability/incapacity
Arm/Group | Intervention: Targeted Infection Control Program | Control
Serious Adverse Events (participants affected / at risk) | 0/203 | 0/215
Other Adverse Events (participants affected / at risk) | 0/203 | 0/215

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No